CLINICAL TRIAL: NCT07333638
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Different Doses of Naltrexone Implant in Patients With Alcohol Use Disorder
Brief Title: Phase II Clinical Study on the Efficacy and Safety of Naltrexone Implant in Patients With Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen Sciencare Medical Industries Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SK2007-NQT-201
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: AUD
Keywords: naltrexone implant
MeSH Terms: interventions — Population Groups; Naltrexone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low-dose group (naltrexone implant 0.9 g ) (Experimental)
  Interventions: Drug: low-dose group (naltrexone implant 0.9 g + general supportive psychological counseling)
- high-dose group (naltrexone implant 1.5 g ) (Experimental)
  Interventions: Drug: high-dose group (naltrexone implant 1.5 g + general supportive psychological counseling)
- control group (placebo ) (Placebo Comparator)
  Interventions: Other: control group (placebo + general supportive psychological counseling)

INTERVENTIONS:
Drug: low-dose group (naltrexone implant 0.9 g + general supportive psychological counseling) — low-dose group (naltrexone implant 0.9 g + general supportive psychological counseling)
  Arms: low-dose group (naltrexone implant 0.9 g )
Drug: high-dose group (naltrexone implant 1.5 g + general supportive psychological counseling) — high-dose group (naltrexone implant 1.5 g + general supportive psychological counseling)
  Arms: high-dose group (naltrexone implant 1.5 g )
Other: control group (placebo + general supportive psychological counseling) — control group (placebo + general supportive psychological counseling)
  Arms: control group (placebo )

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase II clinical trial. The study plans to enroll 210 adult patients with alcohol use disorder. After signing the informed consent form and undergoing screening based on inclusion/exclusion criteria, eligible participants will be randomly assigned to the low-dose group (naltrexone implant 0.9 g + general supportive psychological counseling), high-dose group (naltrexone implant 1.5 g + general supportive psychological counseling), and control group (placebo + general supportive psychological counseling) in a 1:1:1 ratio. On Day 0, participants will receive a single subcutaneous abdominal incision implantation with either 0.9 g or 1.5 g of naltrexone implant or placebo. Efficacy assessment will follow up to 24 weeks after randomization/dosing, while safety assessment will follow up to 48 weeks. There will be a total of 13 follow-up visits. Except for Day 3 (Visit 3) and Week 36 (Visit 12), which are telephone follow-ups, all other visits will be outpatient follow-ups. The first 24 weeks of the study will be double-blind. After completing the Week 24 follow-up, all participants will undergo efficacy assessment. Then they will enter the open-label observation period, followed up until Week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical study; fully understand and are informed about the study and sign the informed consent form; willing and able to comply with and complete all trial procedures; |
2. Age ≥18 years at the time of signing the informed consent form; |
3. Diagnosis of moderate or severe Alcohol Use Disorder based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (meeting four or more diagnostic criteria, see Appendix 1 for details); |
4. Completed detoxification treatment and had no significant alcohol withdrawal symptoms for at least one week (≥7 days) prior to randomization/administration [Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar) score <7 points (see Appendix 2 for specific assessment method)]; |
5. Able to provide Timeline Followback (TLFB) alcohol use information for the 2 weeks during detoxification and/or prior to screening; |
6. Had at least two heavy drinking days per week during the 4 weeks of detoxification and/or prior to screening; |
7. Qualified subjects of childbearing potential (male and female) must agree to use effective contraceptive methods (hormonal or barrier method or abstinence) with their partner during the trial period.

Exclusion Criteria:

1. The investigator judges that participation in this study is not in the best interest of the subject, or any other condition that would make it unsafe for the subject to participate in the study; |
2. Pregnancy, positive pregnancy test for women of childbearing potential, or lactating women, including women of childbearing potential planning to become pregnant during the study period. Note: Women of childbearing potential here refer to women capable of becoming pregnant. Must meet the following criteria, regardless of sexual orientation or tubal ligation: 1) No hysterectomy or bilateral oophorectomy; or 2) Have not been naturally postmenopausal for more than 12 consecutive months (i.e., have had menses at any time in the preceding 12 consecutive months); |
3. Significant abnormal liver function (e.g., AST or ALT >2 times the upper limit of normal) or liver failure [including but not limited to: ascites, prolonged prothrombin time, International Normalized Ratio (INR) ≥1.7, esophageal variceal disease] or hepatobiliary ultrasound shows results that significantly impact the judgment of the study drug's efficacy and safety; |
4. Suffering from clinically uncontrolled active infectious diseases, such as active Hepatitis B [Hepatitis B surface antigen (HBsAg) positive and Hepatitis B virus (HBV) DNA copy number >1000 IU/ml], active Hepatitis C [Hepatitis C virus antibody positive and Hepatitis C virus (HCV)-RNA positive], etc.; |
5. History of congenital bleeding disorders (e.g., hemophilia) or any clinically significant active bleeding, or platelet dysfunction, or prothrombin time (PT) exceeding the upper normal limit by more than 3 seconds, or platelet count <50×10⁹/L; |
6. Previous history of severe pancreatitis or severe delirium tremens;
7. In the investigator's judgment, the subject has any severe/uncontrolled systemic disease (e.g., respiratory, circulatory, digestive, nervous, hematological, urogenital, endocrine systems) or mental illness (e.g., major depressive disorder, schizophrenia, bipolar disorder, etc.) or other major diseases that the investigator believes would prevent providing informed consent, make participation in the study unsafe, complicate the interpretation of study outcome data, or otherwise affect the achievement of study objectives;
8. Likely to require hospitalization or surgery during the study period, including planned elective surgery or hospitalization that cannot be postponed;
9. Diagnosed with substance use disorder (other than alcohol) according to DSM-5 criteria within the current (within one year prior to randomization/administration) period, such as: benzodiazepines, amphetamines, opioids, or cocaine, etc.; |
10. Used medications for relapse prevention (e.g., naltrexone, etc.) or received systematic psychological support therapy within 30 days prior to randomization/administration;
11. Currently receiving treatment for opioid, amphetamine, alcohol, or other substance use disorders, or received opioids within 7 days prior to randomization/administration, likely to require opioid treatment during the study period, or positive urine test for opioids, marijuana, amphetamines, etc., or positive naloxone challenge test on the day of randomization/administration; 12. Allergy to the investigational drug or its excipients (polylactic acid, magnesium stearate), or local anesthetics; |

13. Currently participating in any investigational drug or device study, or used any investigational drug or device within 30 days prior to randomization/administration; 14. Skin infection at the implantation site or systemic skin disease judged to potentially affect the efficacy and safety evaluation of the investigational drug; | 15. Clinical or laboratory evidence of Human Immunodeficiency Virus (HIV) or syphilis carrier/infection. |

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of heavy drinking days during the 24-week observation period post-randomization/treatment | 24-week
  The "Heavy Drinking Days" are divided by the "Days at Risk of Heavy Drinking", with both calculations ending at the cessation of efficacy observation. "Days at Risk of Heavy Drinking" refers to the number of days participants receive efficacy observation during the study. Drinking rates are assessed based on daily alcohol consumption records completed by participants and their families, using the Timeline Follow-Back (TLFB) method. Heavy drinking is defined as "≥5 standard drinks per day for males and ≥4 standard drinks per day for females (In this trial, 1 standard drink = 10 g of pure alcohol).

SECONDARY OUTCOMES:
Change in number of heavy drinking days per month relative to baseline | 24-week
  Specifically, the comparison of total monthly heavy drinking days from randomization/drug administration to the end of follow-up/trial completion with baseline monthly heavy drinking days [calculate monthly corresponding data for weeks 1-24 after randomization/drug administration]; alcohol consumption rate is assessed using the Timeline Follow-Back (TLFB) method based on daily alcohol consumption records completed by subjects and their families . Heavy drinking is defined as "≥5 standard drinks per day for males and ≥4 standard drinks per day for females (in this trial, 1 standard drink = 10 g of pure alcohol).
Alcohol-free days percentage | 24-week
  The "number of alcohol-free days" is divided by the "number of days at risk of alcohol consumption", with both calculations ending at the cessation of efficacy observation. The "number of days at risk of alcohol consumption" is defined as the number of days during which participants receive efficacy observation in the study. According to the Time-Line Follow-Back (TLFB) method, this is calculated based on alcohol consumption records; alcohol consumption is defined as any recorded alcohol consumption behavior, regardless of the quantity or frequency of consumption.
Maximum Consecutive Days of Abstinence | 24-week
  The longest period of continuous alcohol abstinence from randomization/dosing to loss of follow-up/study completion; calculated based on daily alcohol consumption records completed by subjects and their families using the Timeline Follow-Back (TLFB) method.
Daily and Weekly Alcohol Consumption (Daily Drinking Amount and Weekly Total Drinking Amount) | 24-week
  Daily drinking amount and weekly total drinking amount for the corresponding period; calculated based on weekly data from 1 to 24 weeks after randomization/dosing; calculated using the TLFB method based on daily drinking records completed by subjects and their families.
Alcohol Breath Concentration | 24-week
  Random/Post-dosing at 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks; measured by digital alcohol breath tester.
Alcohol Craving Assessment | 24-week
  Randomized/Post-treatment scores at 1 week, 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks; assessed using Visual Analogue Scale (VAS). VAS assessment: One end of the horizontal line is "0", indicating no craving at all; the other end is "10", indicating extreme craving; the middle section represents varying degrees of craving. Participants are asked to select a number from 0-10 that represents their level of craving based on self-perception. The higher the number, the greater the degree of craving.
Alcohol Consequences Score | 24-week
  Randomized/Post-treatment at weeks 4, 8, 12, 16, 20, and 24; assessed using the Alcohol Consequences Checklist
Individual and Social Functioning Status | 24-week
  Assessment of individual and social functioning status at random/4, 8, 12, 16, 20, and 24 weeks post-treatment; Evaluated based on the Personal and Social Performance (PSP) scale:
  A total score of 71-100 indicates no difficulty or only mild difficulty in social functioning and interpersonal relationships A total score of 31-70 indicates varying degrees of impairment in social functioning and interpersonal relationships A total score below 30 indicates poor functioning, requiring active support or close supervision
Follow-up duration (from randomization/dosing to last follow-up) | 24-week
  defined as the time from randomization/dosing to the last follow-up visit.
The proportion of subjects with poor treatment response | 24-week
  defined as the proportion of subjects who were hospitalized for alcohol withdrawal, picked up medication, or lost to follow-up due to poor treatment response;"lost to follow-up due to poor treatment response" is defined as having ≥2 heavy drinking days per week in the 4 weeks prior to loss to follow-up.
Safety assessment indicators | 48-week
  including adverse events (AE) and serious adverse events (SAE) (including local AE and SAE at the implant site), abnormal occurrences of vital signs, physical examination, 12-lead or more ECG, and laboratory safety data (blood routine, urine routine, clinical biochemistry, and coagulation routine) before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University Address: No. 139, Renmin Road Central, Changsha City, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No